CLINICAL TRIAL: NCT02014376
Title: A Phase 2b, Multi-Center, Randomized, Double-Blind, Vehicle-Controlled Study of the Effectiveness and Safety of SD-101 Cream in Subjects With Epidermolysis Bullosa
Brief Title: Study of Effectiveness and Safety of SD-101 in Participants With Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scioderm, Inc. (Industry)
Collaborators: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SD-003
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Epidermolysis Bullosa
Keywords: Epidermolysis Bullosa; Simplex; Recessive Dystrophic; Junctional non-Herlitz; Amicus Therapeutics; Scioderm, Inc.; SD-101 6%; SD-101-6.0; Allantoin 6%; SD-101 3%; SD-101-3.0; Allantoin 3%; Zorblisa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SD-101 Dermal Cream (6%) (Experimental): SD-101 dermal cream (6%) applied topically once daily over the entire body for 90 days.
  Interventions: Drug: SD-101 Dermal Cream (6%)
- SD-101 Dermal Cream (3%) (Experimental): SD-101 dermal cream (3%) applied topically once daily over the entire body for 90 days.
  Interventions: Drug: SD-101 dermal cream (3%)
- Vehicle (0%) (Placebo Comparator): Vehicle dermal cream (SD-101 0%) applied topically once daily over the entire body for 90 days.
  Interventions: Drug: Vehicle (SD-101 0%)

INTERVENTIONS:
Drug: SD-101 dermal cream (3%) — SD-101 is a white, crystalline powder that is formulated within an odorless, soft, white cream base. SD-101-3.0 cream contains allantoin, a diureide glyoxylic acid, at a concentration of 3% and other excipients.
  Other Names: SD-101; SD-101-3.0; Zorblisa
  Arms: SD-101 Dermal Cream (3%)
Drug: SD-101 Dermal Cream (6%) — SD-101 is a white, crystalline powder that is formulated within an odorless, soft, white cream base. SD-101-6.0 cream contains allantoin, a diureide glyoxylic acid, at a concentration of 6% and other excipients.
  Other Names: SD-101; SD-101-6.0; Zorblisa
  Arms: SD-101 Dermal Cream (6%)
Drug: Vehicle (SD-101 0%) — A white, crystalline powder that is formulated within an odorless, soft, white cream base. It contains no allantoin, only excipients.
  Other Names: Placebo Comparator; SD-101-0.0
  Arms: Vehicle (0%)

SUMMARY:
The purpose of this study was to assess whether the topical use of SD-101 cream (3% or 6%) was effective in treating wounds in participants with Simplex, Recessive Dystrophic, or Junctional non-Herlitz Epidermolysis Bullosa (EB).

DETAILED DESCRIPTION:
This was a Phase 2b, multi-center, randomized, double-blind, vehicle-controlled study to assess the efficacy and safety of SD-101 dermal cream (3% or 6%) on skin lesions in participants with Simplex, Recessive Dystrophic, or Junctional non-Herlitz EB.

SD-101 cream [containing 3% or 6% or vehicle (0%)] was applied topically, once a day to the entire body for a period of 90 days. Eligible participants had a target wound assessed at baseline. Selected target wound had to be at least a certain age and within a prespecified size range at study entry. Photographic confirmation of the target wound location was collected at baseline, and the picture saved from the first visit was used to confirm location of the target wound at subsequent visits. The participant returned to the study site at Week 2, Month 1, Month 4, and Month 5 (at 14, 30, 60, and 90 days, respectively) to have the target wound previously identified at baseline re-assessed for the level of healing. In addition, changes in itching, pain, body surface area coverage of blisters and lesions, and scaring of the healed target wound were also assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent form signed by the participant or the participant's legal representative; if the participant is under the age of majority but capable of providing assent, signed assent from the participant.
* Participant (or caretaker) was willing to comply with all protocol requirements.
* Diagnosis of Simplex, Recessive Dystrophic, or Junctional non-Herlitz EB.
* Participants 6 months of age and older.
* Participants had 1 target wound within a prespecified size range at study entry.
* Target wound was at least 21 days or older.

Exclusion Criteria:

* Participants who did not meet all the entry criteria outlined in inclusion criteria.
* Selected target wound had clinical evidence of local infection.
* Use of any investigational drug within 30 days before enrollment.
* Use of immunotherapy or cytotoxic chemotherapy within 60 days before enrollment.
* Use of systemic or topical steroidal therapy within 30 days before enrollment (inhaled steroids and ophthalmic drops containing steroids were allowed).
* Use of systemic antibiotics within 7 days before enrollment.
* Current or former malignancy.
* Arterial or venous disorder resulting in ulcerated wounds.
* Diabetes mellitus.
* Pregnancy or breastfeeding during the study (a urine pregnancy test was performed at screening for female participants of childbearing potential).
* Females of childbearing potential who were not abstinent and not practicing a medically acceptable method of contraception.
* Known history of cardiac, hepatic, or renal disease.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2014-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Amicus Therapeutics
Locations (7):
- United States (7):
  - Palo Alto, California
  - Chicago, Illinois
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Chapel Hill, North Carolina
  - San Antonio, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Started | 15 | 16 | 17
Received at Least 1 Dose of Study Drug (Intent-to-treat (ITT) Population) | 15 | 16 | 17
Completed | 12 | 15 | 17
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population: Participants who provided informed consent, had been randomized, and had received at least 1 application of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%) | Total
Number analyzed (Participants) | 15 | 16 | 17 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.55 (9.189) | 15.32 (15.565) | 11.57 (10.358) | 12.19 (12.029)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 5 | 22
  Male | 6 | 8 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 6 | 17
  Not Hispanic or Latino | 11 | 9 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 11 | 15 | 16 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Epidermolysis Bullosa Subtype [Count of Participants; unit: Participants]
  Simplex | 3 | 4 | 4 | 11
  Recessive Dystrophic | 10 | 9 | 10 | 29
  Junctional non-Herlitz | 2 | 3 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Participants With Documented Complete Closure Of The Target Wound Within 1 Month After Initiation Of Treatment
Description: The ARANZ SilhouetteStar™, a wound imaging, measurement, and documentation system providing accurate wound assessment, was used to measure the target wound at all visits. Information captured included photographic images, quantitative measures, and other target wound assessment data input to the device by the clinician, all obtained with no contact to the participant's skin. Information about the target wound's measurement history was available on this system so that the serial progression of the target wound status could also be calculated and presented.
Time Frame: Baseline to 1 Month
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Number analyzed (Participants) | 15 | 16 | 17
Participants
  Yes | 8 | 6 | 7
  No | 7 | 10 | 10
Statistical Analysis 1: Comparison: SD-101 Dermal Cream (6%) vs Vehicle (0%); Test type: Superiority; p = 0.3699, Fisher Exact

2. Secondary Outcome: Participants With Documented Complete Closure Of The Target Wound Within 2 And 3 Months After Initiation Of Treatment
Description: as for outcome 1
Time Frame: Baseline to Month 2 and Month 3
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Number analyzed (Participants) | 15 | 16 | 17
Participants
  Yes: Month 2 | 9 | 7 | 7
  No: Month 2 | 6 | 9 | 10
  Yes: Month 3 | 9 | 9 | 9
  No: Month 3 | 6 | 7 | 8

3. Secondary Outcome: Percentage Change From Baseline In Lesional Skin Based On Body Surface Area Index (BSAI) Measurements At Month 3
Description: The BSAI is a global measure of disease "spread" with weighting factors. Lesional skin consisted of area(s) that could contain any of the following: blisters, bullae, erosions, ulcerations, scabbing and eschars, as well as areas that are weeping, sloughing, oozing, crusted and denuded. The percentage, ranging from 0% to 100%, of affected body surface area was recorded for each defined body region (head/neck, upper limbs, trunk [includes groin], and lower limbs), multiplied by the weighting factor, and then summed for all body regions to calculate the BSAI. The BSAI affected with blisters and wounds was calculated at baseline and Month 3 to assess the total affected area. Percentage change from baseline was calculated as follows: Percentage change from baseline = 100*(Post-baseline value minus Baseline value) divided by Baseline value. Mean percentage change from baseline in BSAI is reported. Only participants with data available for analysis at the specified time point are presented.
Time Frame: Baseline, Month 3
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of BSAI
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Number analyzed (Participants) | 12 | 15 | 17
percentage of BSAI | -28.02 (35.949) | -42.52 (37.624) | -5.75 (110.470)

4. Secondary Outcome: Participants Experiencing A Change From Baseline In Itching At Day 7
Description: The Itch Man Pruritus Assessment Tool was used to measure the intensity of itching. Itching was assessed and reported at Baseline and Day 7. For participants 6 months to 5 years of age, itching was assessed using the caretaker's response, while in participants 6 years and older, itching was self-reported.
Time Frame: Baseline, Day 7
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Number analyzed (Participants) | 15 | 16 | 17
Participants
  Improved | 5 | 4 | 7
  Not Improved | 9 | 12 | 10
  Missing | 1 | 0 | 0

5. Secondary Outcome: Change From Baseline In Pain At Day 7
Description: Pain was assessed at Baseline and Day 7. The presence and intensity of pain was assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) Pain Scale for participants 6 months to 3 years of age. For participants aged 4 years and older, the Wong Faces Pain Scale was used. Scores were attributed for each of the 5 categories in the FLACC scale from 0 to 2, which resulted in a total score between 0 and 10. The Wong Faces Pain scale used 1 item to rate pain on a 0 to 10 scale. Higher score values indicated more pain.
Time Frame: Baseline, Day 7
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Number analyzed (Participants) | 15 | 16 | 17
score on a scale
  FLACC Pain Scale: number analyzed (Participants) | 2 | 6 | 5
  FLACC Pain Scale | 0.50 (0.707) | -0.17 (5.307) | -1.60 (2.881)
  Wong Faces Pain Scale: number analyzed (Participants) | 11 | 10 | 12
  Wong Faces Pain Scale | 0.91 (2.119) | -0.70 (2.908) | 1.08 (2.353)

6. Secondary Outcome: Participants With Scarring At Week 2, Month 1, Month 2, And Month 3
Description: In the event of a healed wound, where complete closure was confirmed, the extent of scarring was assessed as "Present" or "Absent" at all post-baseline visits (Week 2 and Months 1, 2, and 3).
Time Frame: Week 2, Month 1, Month 2, and Month 3
Population: Intent-to-treat (ITT) Population: Participants who provided informed consent, had been randomized, had received at least 1 application of study drug, and whose target wounds healed while receiving study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
Number analyzed (Participants) | 9 | 9 | 9
Participants
  Week 2: number analyzed (Participants) | 4 | 1 | 2
  Week 2: Present | 0 | 0 | 0
  Week 2: Absent | 4 | 1 | 2
  Month 1: number analyzed (Participants) | 4 | 5 | 5
  Month 1: Present | 2 | 2 | 2
  Month 1: Absent | 2 | 3 | 3
  Month 2: number analyzed (Participants) | 1 | 1 | 0
  Month 2: Present | 0 | 1 | 0
  Month 2: Absent | 1 | 0 | 0
  Month 3: number analyzed (Participants) | 0 | 2 | 2
  Month 3: Present | 0 | 0 | 0
  Month 3: Absent | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: From baseline (Day 0) to 30 days after last application of study drug (up to a maximum of 4 months).
Arm/Group | SD-101 Dermal Cream (6%) | SD-101 Dermal Cream (3%) | Vehicle (0%)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/16 | 1/17
Other Adverse Events (participants affected / at risk) | 9/15 | 13/16 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD-101 Dermal Cream (6%) (N=15) | SD-101 Dermal Cream (3%) (N=16) | Vehicle (0%) (N=17)
Bacterial tracheitis (Infections and infestations) | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD-101 Dermal Cream (6%) (N=15) | SD-101 Dermal Cream (3%) (N=16) | Vehicle (0%) (N=17)
Nasopharyngitis (Infections and infestations) | 1 | 4 | 2
Otitis media (Infections and infestations) | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 3 | 2
Application site pain (General disorders) | 2 | 3 | 1
Pain (General disorders) | 2 | 0 | 0
Application site discharge (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2
Aphonia (Nervous system disorders) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Corneal disorder (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Protein deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days